CLINICAL TRIAL: NCT00251017
Title: Impact of Polymorphisms of OAT1, OAT3, and OCT2 on Transportation of Potential Nephrotoxic Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9361701301; DOH94-td-d-113-035(2) (Other Grant/Funding Number: Department of Health, Taiwan)
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Adverse Effects
Keywords: single nucleotide polymorphisms (SNPs); personalized medicines; Subjects 16 years of age or older, of either sex.; Subjects have a medication including vancomycin
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin (Active Comparator): Effects of OCT2 genetic variation in renal elimination of Vancomycin
  Interventions: Procedure: Vancomycin; Procedure: DNA are extracted from the whole blood of subjects

INTERVENTIONS:
Procedure: Vancomycin — Two hour creatinine clearance before and after vancomycin
Procedure: DNA are extracted from the whole blood of subjects

SUMMARY:
Transporters in kidney are critical in detoxification and elimination of xenobiotics from systemic circulation, and thus are major determinants of drug response and sensitivity. Transporters in the renal epithelium control the exposure of renal cells to nephrotoxic drugs and environmental toxins and thus determine xenobiotic-induced nephrotoxicity. Organic anion transporters (OATs) and organic cation transporters (OCTs) are two major classes of secretory transporters in the mammalian kidney. Among the uptake transporters, OAT1, OAT3, or OCT2 appear to be particularly important in the renal basolateral membrane to transport a large variety of endogenous and therapeutic compounds.

Recently, rapid advances in single nucleotide polymorphisms (SNPs) mapping can now be applied to characterize the individual patients who suffer adverse effects to a drug, or those for whom a drug shows efficacy. The aim of this study was to identify and functionally characterize OCT2 variants as a first step towards understanding whether genetic variation in OCT2 may contribute to interindividual differences in renal elimination of vancomycin. Taiwanese patients will be screened and 12 coding region variants of OCT2 will be identified. The non-synonymous variants of OAT1, OAT3, or OCT2 will then be constructed and characterized using in vitro human renal cell models. It is to establish whether genetic variants in OAT1, OAT3, or OCT2 are likely significant contributors to intersubject variability in drug response. In addition, approaches toward prevention of some drug-induced nephrotoxicity are discussed, based on molecular mechanisms of renal accumulation of these drugs. Perhaps the researchers' understanding of OAT1, OAT3, or OCT2 in pharmacogenomics may contribute to the goal of individualized drug therapy. Development of new strategies based on the understanding of their cellular handing may achieve safer and more effective therapy for personalized medicines.

DETAILED DESCRIPTION:
Beta-lactam antibiotics, aminoglycosides, amphotericin B, cyclosporine, nonsteroidal anti-inflammatory drugs, antineoplastic, or antivirus drugs that are used extensively in clinical settings bear the risk of nephrotoxicity. This side effect is dose-dependent and has been attributed mainly to the accumulation of drugs in the renal proximal tubule. When assessing nephrotoxicity, both the dosage and the tubular secretion system, which allows transport of drug from blood to urine via the tubular cells, are important factors. This study was designed to investigate how renal transporters work in the renal secretion of specific drugs.

Transporters in kidney are critical in detoxification and elimination of xenobiotics from systemic circulation, and thus are major determinants of drug response and sensitivity. Transporters in the renal epithelium control the exposure of renal cells to nephrotoxic drugs and environmental toxins and thus determine xenobiotic-induced nephrotoxicity. Organic anion transporters (OATs) and organic cation transporters (OCTs) are two major classes of secretory transporters in the mammalian kidney. Among the uptake transporters, OAT1, OAT3, or OCT2 appear to be particularly important in the renal basolateral membrane to transport a large variety of endogenous and therapeutic compounds.

Recently, rapid advances in single nucleotide polymorphisms (SNPs) mapping can now be applied to characterize the individual patients who suffer adverse effects to a drug, or those for whom a drug shows efficacy. The aim of this study was to identify and functionally characterize OCT2 variants as a first step towards understanding whether genetic variation in OCT2 may contribute to interindividual differences in renal elimination of vancomycin. Taiwanese patients will be screened and 12 coding region variants of OCT2 will be identified. The non-synonymous variants of OAT1, OAT3, or OCT2 will then be constructed and characterized using in vitro human renal cell models. It is to establish whether genetic variants in OAT1, OAT3, or OCT2 are likely significant contributors to intersubject variability in drug response. In addition, approaches toward the prevention of some drug-induced nephrotoxicity are discussed, base on molecular mechanisms of renal accumulation of these drugs. Perhaps our understanding of OAT1, OAT3, or OCT2 in pharmacogenomics may contribute to the goal of individualized drug therapy. Development of new strategies based on the understanding of their cellular handing may achieve safer and more effective therapy for personalized medicines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 16 years of age or older, of either sex.
* Subjects have a medication including vancomycin
* Subjects have realistic expectations of the benefit and limitation of the augmentation procedure, as determined by a willingness to sign the informed consent form after it has been carefully explained.

Exclusion Criteria:

* Subjects have a medical condition that increased the risks of study participation (including pregnancy and poor renal function)
* Subjects are taking medications (nephrotoxicants) that could confound study results.
* Subjects presenting with history of autoimmune disorder, septic shock, or multiple organ failure.
* Subjects with renal failure undergoing dialysis (hemodialysis [HD] or continuous ambulatory peritoneal dialysis [CAPD]), continuous venovenous hemofiltration (CVVH), or continuous arteriovenous hemodiafiltration (CAVHDF).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Single nucleotide polymorphism (SNP), plasma creatinine and vancomycin concentration | 0, 2 hour after Vancomycin administration

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Wang Chern, Ph.D., Study Chair — National Taiwan University; Wen-Je Ko, M.D, Ph.D, Principal Investigator — National Taiwan University Hospital; Fe-Lin Lin, Ph.D., Principal Investigator — National of University; Chiung-Hua Huang, M.S, Study Director — National Taiwan University
Locations (1):
- Department of Surgery, National Taiwan University Hospital, Taipei, Taiwan